CLINICAL TRIAL: NCT05730023
Title: A Multimodal Approach for Clinical Diagnosis and Treatment of Primary Progressive Aphasia, MAINSTREAM ID:3430931
Acronym: MAINSTREAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Collaborators: Fondazione Regionale per la Ricerca Biomedica (Other); Fondazione Mondino (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); IRCCS Fondazione Don Carlo Gnocchi - ONLUS, Milan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MAINSTREAM ID:3430931
Record Dates: First submitted 2023-01-31; First posted 2023-02-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Primary Progressive Aphasia
Keywords: Behavioral and neural effects of tDCS combined with language training; Alzheimer's disease and other dementias
MeSH Terms: conditions — Aphasia, Primary Progressive; Behavior; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active tDCS plus individualized language training (Experimental): The group will receive five consecutive days a week for two weeks of 25 minutes sessions of Active tDCS combined with an individualized language training
  Interventions: Device: Active tDCS; Behavioral: individualized language training
- Placebo tDCS plus individualized language training (Active Comparator): The group will receive five consecutive days a week for two weeks of 25 minutes sessions of Placebo tDCS combined with an individualized language training
  Interventions: Behavioral: individualized language training; Device: Placebo tDCS

INTERVENTIONS:
Device: Active tDCS — Active tDCS (anode will be applied over the left DLPFC with the cathode over the right supraorbital region);
  Arms: Active tDCS plus individualized language training
Behavioral: individualized language training — individualized language training
Device: Placebo tDCS — Placebo tDCS (the current will be turned off 10 seconds after the beginning and turned on for the last 10 seconds of the stimulation period);
  Arms: Placebo tDCS plus individualized language training

SUMMARY:
Primary Progressive Aphasia (PPA) is a syndrome due to different neurodegenerative disorders selectively disrupting language functions. PPA specialist care is underdeveloped. There are very few specialists (neurologists, psychiatrists, neuropsychologists and speech therapists) and few hospitals- or community-based services dedicated to diagnosis and continuing care. Currently, healthcare systems struggle to provide adequate coverage of diagnostic services, and care is too often fragmented, uncoordinated, and unresponsive to the needs of people with PPA and their families. Recently attention has been gained by digital-health technologies, such immunoassay analyzer and high-field MRI, the most promising approaches to increase our understanding of neurodegeneration, and by new non-invasive brain stimulation techniques such as transcranial direct current stimulation (tDCS) that allow a personalized treatment approach. Our goal is to develop a new treatment approach in PPA in which the regional secondary care centers participating in this project should be the hub of a regional network. The MAINSTREAM (WP2- Efficacy of personalized training in the early stage of PPA) looks forward to introduce and evaluate therapeutic innovation such as tDCS coupled with language therapy in rehabilitation settings (WP2 Early Treatment).

This objective will be pursued by conducting a randomized controlled pilot study in order to evaluate the efficacy of a combined treatment of Active (anodal) tDCS and individualized language training compared to Placebo tDCS combined with individualized language training in a subgroup of mild PPA defined using the Progressive Aphasia Severity Scale (PASS) (Sapolsky D, Domoto-Reilly K, Dickerson BCJA. Use of the Progressive Aphasia Severity Scale (PASS) in Monitoring Speech and Language Status in PPA. (2014) 28(8-9):993-1003).

DETAILED DESCRIPTION:
60 patients with PPA will be recruited from IRCCS Istituto Centro San Giovanni di Dio, Fatebenefratelli, Brescia; IRCCS Fondazione Istituto Neurologico Nazionale C. Mondino, Pavia; Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan and Fondazione Don Carlo Gnocchi - ONLUS, Milan.

The diagnostic evaluation will include cognitive and language testing, neurologic examination and neuroimaging (Magnetic Resonance Imaging (MRI) or Positron Emission Tomography PET)).

All the patients will undergo five consecutive days a week for two weeks of treatment sessions of 25 minutes:

* 30 patients will receive Active tDCS over dorsolateral prefrontal cortex-DLPFC (anode over the left DLPFC with the cathode over the right supraorbital region) while performing an individualized language training;
* 30 patients will receive Placebo tDCS during an individualized language training.

The two groups will be matched for sex, age, education, language severity (as defined in the Frontotemporal Dementia Clinical Dementia Rating subscale), and overall severity according to the FTD Clinical Dementia Rating.

Two trained neuropsychologists will administer the neuropsychological testing at baseline (T0), post-treatment (T1) and 3-months (T2) follow-up. All of assessments will be conducted by the same assessor.

To elucidate the mechanisms underlying tDCS effects, Magnetic Resonance Imaging (MRI) and bimolecular data will be collected at T0 and T1 (after the treatment).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis PPA according to the current clinical criteria (Gorno-Tempini et al., 2011);
* Mild PPA defined using the Progressive Aphasia Severity Scale (PASS);
* Italian native speakers.

Exclusion Criteria:

* Presence of developmental disorders;
* Presence of any medical or psychiatric illness that could interfere in completing assessments;
* Presence of any medical condition that represents a contraindication to tDCS.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in measure of naming as assessed by International Picture Naming Project Task (IPNP) | Baseline up to 2 weeks and 3 months
  International Picture Naming Project Task (IPNP): trained (score range: min= 0, max= 32, higher score=better outcome) and untrained object items (score range: min= 0, max= 32, higher score=better outcome); action items (score range: min= 0, max= 60, higher score=better outcome).

SECONDARY OUTCOMES:
Change in measure of quality of life as assessed by Stroke and Aphasia Quality of Life Scale - 39 (SAQoL-39) | Baseline up to 2 weeks and 3 months
  Stroke and Aphasia Quality of Life Scale - 39 (SAQoL-39) is a measure of health-related quality of life in people with long-term aphasia. It provides a total score from 1 to 5 (higher score=better outcome) and it analyzes the following four domains: physical (score range: min= 1, max= 5, higher score=better outcome); psychosocial (score range: min= 1, max= 5, higher score=better outcome); communication (score range: min= 1, max= 5, higher score=better outcome) and energy (score range: min= 1, max= 5, higher score=better outcome).
Change in measure of quality of life as assessed by Communication Outcome After Stroke (COAST) | Baseline up to 2 weeks and 3 months
  Communication Outcome After Stroke (COAST) is a measure of the functional communication in daily activities and of the impact of the quality of life point of view of aphasia patient (COAST total score range: min= 0, max= 80, higher score=better outcome) and their carer (Carer COAST total score range: min= 0, max= 80, higher score=better outcome).
Change in measure of quality of life as assessed by Functional Outcome Questionnaire-aphasia | Baseline up to 2 weeks and 3 months
  Functional Outcome Questionnaire-aphasia is a measure of aphasia's functional and pragmatic communication in home and community settings, It provides a total score from 32 to 160 (higher score=better outcome) and it is divided into four subscales: communicating basic needs (CBN score range: min= 1, max= 35, higher score=better outcome); making routine requests (MRR score range: min= 1, max= 35, higher score=better outcome); communicating new information (CNI score range: min= 1, max= 40, higher score=better outcome) and attention/other communication skills (AO score range: min= 1, max= 50, higher score=better outcome).
Change in dementia severity as assessed by Frontotemporal Dementia- Clinical Dementia Rating Scale (FTD-CDR)- Sum of Boxes | Baseline up to 2 weeks and 3 months
  Frontotemporal Dementia- Clinical Dementia Rating Scale (FTD-CDR)- Sum of Boxes (score range: min= 0, max= 24, higher score=worse outcome).
Change in dementia severity as assessed by Global Clinical Dementia Rating (CDR) plus NACC FTLD | Baseline up to 2 weeks and 3 months
  Global Clinical Dementia Rating (CDR) plus NACC FTLD (score range: min= 0, max= 3, higher score=worse outcome).
Change in aphasia severity as assessed by Progressive Aphasia Severity Scale (PASS) | Baseline up to 2 weeks and 3 months
  PASS is a measure of severity and progression of language deficits in patients with PPA. The scale assesses ten linguistic domains (each score range: min= 0, max= 3): articulation (higher score=worse outcome), fluency (higher score=worse outcome), syntax and grammar (higher score=worse outcome), word retrieval and expression (higher score=worse outcome), repetition (higher score=worse outcome), auditory comprehension (higher score=worse outcome), single word comprehension (higher score=worse outcome), reading (higher score=worse outcome), writing (higher score=worse outcome) and functional communication (higher score=worse outcome). Moreover, it analyzes three supplemental domains (each score range: min= 0, max= 3): initiation of conversation (higher score=worse outcome), turn taking during conversation (higher score=worse outcome) and generation of language (higher score=worse outcome).
Change in functional communication skills as assessed by Lincoln Speech Questionnaire | Baseline up to 2 weeks and 3 months
  Lincoln Speech Questionnaire provides a speech score (score range: min= 0, max= 14, higher score=better outcome) and an understanding score (score range: min= 0, max= 5, higher score=better outcome).
Change in aphasia severity as assessed by Communication Severity Rating Scale (Goodglass and Kaplan) | Baseline up to 2 weeks and 3 months
  Communication Severity Rating Scale (Goodglass and Kaplan): score range: min= 0, max= 5, higher score=better outcome.
Change in depressive symptoms as assessed by Beck Depression Inventory (BDI) | Baseline up to 2 weeks and 3 months
  Beck Depression Inventory (BDI): score range: min= 0, max= 63, higher score=worse outcome
Change in behavior and personality as assessed by Frontal Behavioral Inventory (FBI) | Baseline up to 2 weeks and 3 months
  Frontal Behavioral Inventory (FBI): score range: min= 0, max= 72, higher score=worse outcome.
Change in measure of naming as assessed by Picture Naming subtest from Screening for Aphasia in NeuroDegeneration (SAND) | Baseline up to 2 weeks and 3 months
  Picture Naming subtest from Screening for Aphasia in NeuroDegeneration (SAND) provides total score (score range: min= 0, max= 14, higher score=better outcome), living score (score range: min= 0, max= 7, higher score=better outcome) and non-living score (score range: min= 0, max= 7, higher score=better outcome).
Change in measure of comprehension as assessed by Auditory sentence comprehension subtest from Screening for Aphasia in NeuroDegeneration (SAND) | Baseline up to 2 weeks and 3 months
  Auditory sentence comprehension subtest from Screening for Aphasia in NeuroDegeneration (SAND): total score range: min= 0, max= 8, higher score=better outcome.
Change in measure of comprehension as assessed by Single-word comprehension subtest from Screening for Aphasia in NeuroDegeneration (SAND) | Baseline up to 2 weeks and 3 months
  Single-word comprehension subtest from Screening for Aphasia in NeuroDegeneration (SAND) provides total score (score range: min= 0, max= 12, higher score=better outcome), living score (score range: min= 0, max= 6, higher score=better outcome) and non-living score (score range: min= 0, max= 6, higher score=better outcome).
Change in measure of repetition as assessed by Repetition subtest from Screening for Aphasia in NeuroDegeneration (SAND) | Baseline up to 2 weeks and 3 months
  Repetition subtest from Screening for Aphasia in NeuroDegeneration (SAND) provides total score (score range: min= 0, max= 10, higher score=better outcome), words score (score range: min= 0, max= 6, higher score=better outcome) and non-words score (score range: min= 0, max= 4, higher score=better outcome).
Change in measure of repetition as assessed by Sentence repetition subtest from Screening for Aphasia in NeuroDegeneration (SAND) | Baseline up to 2 weeks and 3 months
  Sentence repetition subtest from Screening for Aphasia in NeuroDegeneration (SAND) provides total score (score range: min= 0, max= 6, higher score=better outcome), predictable sentences score (score range: min= 0, max= 3, higher score=better outcome) and unpredictable sentences score (score range: min= 0, max= 3, higher score=better outcome).
Change in measure of reading as assessed by Reading subtest from Screening for Aphasia in NeuroDegeneration (SAND) | Baseline up to 2 weeks and 3 months
  Reading subtest from Screening for Aphasia in NeuroDegeneration (SAND) provides total score (score range: min= 0, max= 16, higher score=better outcome), words score (score range: min= 0, max= 12, higher score=better outcome) and non-words score (score range: min= 0, max= 4, higher score=better outcome).
Change in measure of writing as assessed by Writing subtest from Screening for Aphasia in NeuroDegeneration (SAND) | Baseline up to 2 weeks and 3 months
  Writing subtest from Screening for Aphasia in NeuroDegeneration (SAND) provides Information Units score (score range: min= 0, max= 6, higher score=better outcome), total number of words score (score range: min= 0, max= no limits, higher score=better outcome), number of nouns/total number of words score (score range: min= 0, max= 1, higher score=better outcome), number of verbs/total number of words (score range: min= 0, max= 1, higher score=better outcome), number of correct syntactic structures/total number of syntactic structures score (score range: min= 0, max= 1, higher score=better outcome), number of orthographic errors score (score range: min= 0, max= no limits, higher score=worse outcome), number of lexico-semantic errors/number of words score (score range: min= 0, max= 1, higher score=worse outcome).
Change in measure of semantics as assessed by Semantic association subtest from Screening for Aphasia in NeuroDegeneration (SAND) | Baseline up to 2 weeks and 3 months
  Semantic association subtest from Screening for Aphasia in NeuroDegeneration (SAND): total score range: min= 0, max= 4, higher score=better outcome.
Change in measure of oral production as assessed by Picture description subtest from Screening for Aphasia in NeuroDegeneration (SAND) | Baseline up to 2 weeks and 3 months
  Picture description subtest from SAND provides Information Units score (score range: min= 0, max= 8, higher score=better outcome), total number of words score (score range: min= 0, max= no limits, higher score=better outcome), number of nouns/total number of words score (score range: min= 0, max= 1, higher score=better outcome), number of verbs/total number of words score (score range: min= 0, max= 1, higher score=better outcome), number of sentences score (score range: min= 0, max= no limits, higher score=better outcome), number of subordinates/number of sentences score (score range: min= 0, max= no limits, higher score=better outcome), number of repaired sequences/number of words score (score range: min= 0, max= 1, higher score=worse outcome), number of phonological errors/number of words (score range: min= 0, max= 1, higher score=worse outcome), number of lexico-semantic errors/number of words (score range: min= 0, max= 1, higher score=worse outcome).
Change in measure of naming as assessed by Subtest from Aachener Aphasie Test (AAT) | Baseline up to 2 weeks and 3 months
  Naming subtest from Aachener Aphasie Test (AAT): score range: min= 0, max= 120, higher score=better outcome.
Change in measure of object naming as assessed by Subtest from Battery for the Assessment of Aphasic Disorders (BADA) | Baseline up to 2 weeks and 3 months
  Subtest from Battery for the Assessment of Aphasic Disorders (BADA): score range: min= 0, max= 30, higher score=better outcome.
Change in measure of fluency abilities as assessed by Verbal Fluency (semantic and phonemic) | Baseline up to 2 weeks and 3 months
  Verbal Fluency (semantic and phonemic): score range min= 0, max= no limits, higher score=better outcome.
Change in measure of constructional praxia as assessed by Rey-Osterrieth Complex Figure-Copy | Baseline up to 2 weeks and 3 months
  Rey-Osterrieth Complex Figure-Copy: score range min= 0, max= 36, higher score=better outcome.
Change in measure of verbal long-term memory as assessed by Story Recall | Baseline up to 2 weeks and 3 months
  Story Recall: score range min= 0, max= 28, higher score=better outcome.
Change in measure of nonverbal long-term memory as assessed by Rey-Osterrieth Complex Figure-Recall | Baseline up to 2 weeks and 3 months
  Rey-Osterrieth Complex Figure-Recall: score range min= 0, max= 36, higher score=better outcome.
Change in measure of attentional abilities as assessed by Trial Making Test | Baseline up to 2 weeks and 3 months
  Trial Making Test: score range: min= n/a, max= no limits, higher score=worse outcome.
Change in measure of executive abilities as assessed by Stroop Test | Baseline up to 2 weeks and 3 months
  Stroop Test: score range: min= n/a, max= no limits, higher score=worse outcome.
Change in measure of global cognitive impairment as assessed by Mini Mental State Examination (MMSE) | Baseline up to 2 weeks and 3 months
  Mini Mental State Examination (MMSE): score range: min= 0, max= 30, higher score=better outcome.
Change in molecular biomarkers as assessed by the size and the concentration of plasma Extracellular vesicles (EVs) | Baseline up to 2 weeks
  Size and the concentration of plasma EVs
Change in molecular biomarkers as assessed by Neurofilament light chain (NFL) levels | Baseline up to 2 weeks
  Neurofilament light chain (NFL) levels
Change in molecular biomarkers as assessed by Glial Fibrillary Acidic Protein (GFAP) levels | Baseline up to 2 weeks
  Glial Fibrillary Acidic Protein (GFAP) levels
Change in molecular biomarkers as assessed by brain-derived neurotrophic factor (BDNF) | Baseline up to 2 weeks
  Brain-derived neurotrophic factor (BDNF) levels
Change in molecular biomarkers as assessed by neurogranin levels | Baseline up to 2 weeks
  Neurogranin levels
Change in functional connectivity as derived from resting-state functional MRI | Baseline up to 2 weeks
  Functional connectivity as derived from resting-state functional MRI
Change in structural connectivity as derived from diffusion-weighted MRI | Baseline up to 2 weeks
  Structural connectivity as derived from diffusion-weighted MRI

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cotelli, Principal Investigator — IRCCS Istituto Centro San Giovanni di Dio- Fatebenefratelli
Locations (4):
- Italy (4):
  - Maria Cotelli, Brescia, BS
  - Tiziana Carandini, Milan, MI
  - Francesca Baglio, Milan, MI
  - Stefano F. Cappa, Pavia, PV

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cotelli M, Baglio F, Manenti R, Blasi V, Galimberti D, Gobbi E, Pagnoni I, Rossetto F, Rotondo E, Esposito V, De Icco R, Giudice C, Tassorelli C, Catricala E, Perini G, Alaimo C, Campana E, Benussi L, Ghidoni R, Binetti G, Carandini T, Cappa SF. A Multimodal Approach for Clinical Diagnosis and Treatment of Primary Progressive Aphasia (MAINSTREAM): A Study Protocol. Brain Sci. 2023 Jul 12;13(7):1060. doi: 10.3390/brainsci13071060. PMID 37508992